CLINICAL TRIAL: NCT05629260
Title: A Multi-center, Prospective Study of Clinical Outcome and Immune Reconstruction in G-CSF/ATG and PT-Cy Based Haploidentical Transplantation
Brief Title: The Optimization of Haploidentical Hematopoietic Stem Cell Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Other Study IDs: GM-2021-13560
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Hematological Malignancy
Keywords: Haploidentical Transplantation; G-CSF/ATG; PT-Cy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- G-CSF/ATG group: Patients in the G-CSF/ATG group received a modified Bu/Cy plus ATG conditioning regimen as follows: cytarabine (4/g m2 per day IV.) on days -10 to -9; Bu (3.2 mg/kg per day IV.) on days -8 to -6; Cy (1.8 g/m2 per day IV.) on days -5 to -4; methyl chloride hexamethylene urea nitrate (Me-CCNU) (250 mg/m2 per day orally) once on day -3; and ATG (2.5 mg/kg per day IV; rabbit, Sang Stat, Lyon, France) on days -5 to -2.
  Interventions: Drug: ATG
- PT-Cy group: Patients in PT-Cy group received a Bu/Flu/Cy-based conditioning regimen as follows: Flu (40 mg/m2 or 1 mg/kg IV) on days -8 to -4; Bu (3.2 mg kg/ d-1 IV) on days -7 to -4; Cy (14.5-40 mg/kg IV) on days -3 to -2;±cytarabine (3 g/m2/d IV) on days -9 to -8; and ± IDA (15 mg/m2/d IV) on days -9 to -8. The addition of IDA and/or cytarabine depended on the performance status of the patients and whether the patients were in relapse status. High-dose PTCy (50 mg/kg/d IV) was administered on days +3 and +4.
  Interventions: Drug: Post-transplantation cyclophosphamide

INTERVENTIONS:
Drug: ATG — Patients with intermediate-high risk hematologic malignancy who are indicated for allogeneic hematopoietic stem cell transplantation (allo-HSCT) and absence of HLA matched donors will be treated with haplo-HSCT, with G-CSF/ATG based protocol.
  Groups: G-CSF/ATG group
Drug: Post-transplantation cyclophosphamide — Patients with intermediate-high risk hematologic malignancy who are indicated for allogeneic hematopoietic stem cell transplantation (allo-HSCT) and absence of HLA matched donors will be treated with haplo-HSCT with PT-Cy based protocol.
  Groups: PT-Cy group

SUMMARY:
The goal of this observational study is to compare the incidence of relapse in G-CSF/ATG based and PT-Cy based haploidentical transplantation] in [patients aged 18 to 55 years with a diagnosis of hematological malignancies who unmanipulated haplo-HSCT with myeloablative conditioning]. The main question it aims to answer are:

Primary objective: To compare the incidence of relapse in G-CSF/ATG based and PT-Cy based haploidentical transplantation and illustrate the possible immune mechanism.

Secondary objectives: To compare CMV infection, GVHD and survival outcomes, and to observe the dynamic immune reconstitution of G-CSF/ATG based or PT-Cy based model.

Exploratory objectives: To compare the long-term quality of life among recipients who receive G-CSF/ATG based or PT-Cy based protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed as acute leukemia with transplant indications in ≤ CR2;
2. Lack of available, HLA-identical, related sibling or unrelated donor;
3. Female or male, age: 18-55 years old;
4. ECOG performance status 0-2;
5. Adequate organ function as defined by the following criteria:

   Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤2.5× upper limit of normal (ULN), or AST and ALT ≤5× ULN if liver function abnormalities are due to underlying malignancy Total serum bilirubin≤1.5× ULN Serum creatinine≤2.5× ULN
6. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment;
7. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Uncontrollable active infection;
2. Severe organic impairment: hepatic and renal impairment;
3. Any of the following within 6 months prior to starting study treatment: myocardial infarction, severe/unstable angina, congestive heart failure, or cerebrovascular accident including transient ischemic attack;
4. Pregnancy or breastfeeding;
5. Psychiatric disorders;
6. Don't sign the informed consent;
7. Prior/concurrent clinical study experience;
8. Other conditions:

   * Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
   * Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals (in conjunction with section 1.61 of the ICH-GCP Ordinance E6)
   * Any specific situation during study implementation/course that may rise ethics considerations
   * Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with hematologic malignancy who are indicated for allogeneic hematopoietic stem cell transplantation (allo-HSCT) and absence of HLA matched donors will be treated with haplo-HSCT with either G-CSF/ATG based or PT-Cy based protocols（4:1）
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with disease relapse | 1 year
  The cumulative incidence of relapse of the primary disease.

SECONDARY OUTCOMES:
Incidence of CMV disease | 6 months
  The cumulative incidences of CMV disease in participants after transplantation
Cumulative incidences of aGVHD | 100 days
  The diagnosis and grading of aGVHD are based on the modified Glucksberg grading standard.
Cumulative incidences of cGVHD | 1 year
  Chronic GVHD can be classified as "limited" or "extensive" according to the Seattle criteria, and also be classified as "mild" or "moderate" or "severe" according to the National Institutes of Health (NIH) criteria.
Percent of participants with overall survival | 1 year
  Overall survival (OS) is defined as the time from randomization to death resulting from any cause.
Dynamic immune reconstitution | 1 year
  The main immune cell subsets include: T cell, B cell, NK cell, and Monocytes
Neutrophil engraftment | 1 month
  Neutrophil engraftment is defined as the first of 3 consecutive days with an absolute neutrophil count > 0.5 × 10^9/L.
Platelet engraftment | 1 month
  Platelet engraftment is defined as the first of 7 consecutive days with an absolute platelet count > 20 × 10^9/L independent from transfusion
Transplantation-related mortality | 1 year
  Death due to causes unrelated to the underlying disease

CONTACTS AND LOCATIONS:
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided